CLINICAL TRIAL: NCT04739475
Title: Association of Stress and Non-surgical Periodontal Therapy (NPT) Outcome in Patients With Periodontitis Stage III/V Grade A/B Generalised
Brief Title: Effect of Stress on Periodontal Therapy (NPT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Giacomo Baima, Principal investigator, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTurin01
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Stress, Psychological; Periodontal Diseases; Periodontitis; Non Surgical Periodontal Therapy; Inflammation; Bleeding on Probing
MeSH Terms: conditions — Stress, Psychological; Periodontal Diseases; Periodontitis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non surgical Periodontal Therapy NPT (Other): Conventional staging debridement (CSD) according to the severity of periodontal disease in 2 to 4 appointments at day 0, 7, 14 and 21.
  Supra and subgingival scaling and polishing will be performed by the use of manual and ultrasonic instruments and oral hygiene instructions will be given. Patients will be instructed to use interdental brushes with appropriate size interdental brushes or dental floss when interdental embrasures will not allow for interdental brushing.
  Interventions: Procedure: Non Surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Non Surgical Periodontal Therapy — Conventional staging debridement (CSD) according to the severity of periodontal disease in 2 to 4 appointments at day 0, 7, 14 and 21.
  Supra and subgingival scaling and polishing will be performed by the use of manual and ultrasonic instruments and oral hygiene instructions will be given. Patients will be instructed to use interdental brushes with appropriate size interdental brushes or dental floss when interdental embrasures will not allow for interdental brushing.

SUMMARY:
Aim of this study:

is to evaluate the influence of stress level on the response of non surgical periodontal therapy in patients affected by severe periodontitis divided into "Medium/High stress level" or "Low stress level" based on the Perceived Stress Scale (PSS). The defined primary outcome referring to the clinical response of the patients is the bleeding index, Full-Mouth Bleeding Score (FMBS), as a clinical sign of inflammation.

Materials and Methods:

Monocentric prospective triple blinded study. A single evaluator conducting all the psychologic tests, a single operator blinded to the results of the psychologic tests doing all the clinical measurements, and the patients will be initially blinded to the category of stress that they'll belong to. The minimum number of patients to enrol will be 89 based on a sample calculation.

Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

Age from 20 to 80 years Diagnosis of Periodontitis stage III/IV according to the new classification (2018); Presence of at least 14 teeth, with a minimum of 10 sites with PD at least > 5 mm and radiographic evidence of alveolar bone loss.

Written informed consent

Exclusion Criteria.

The presence of any of the following will exclude a subject from study enrollment:

Smokers > 10 cig/die Patients with orthodontic appliances; Pregnant or lactating women; Individuals who have received periodontal treatment in the 6 months prior to recruitment; Patients with systemic diseases that could interfere the clinical response to periodontal treatment (i.e. diabetes); Subjects under treatment with antibiotics, steroidal and/or non-steroidal anti-inflammatory medication 3 weeks prior to the visit and patients treated with antiepileptic drugs

Operative procedure:

Clinical parameters and psychologic test will be done at the baseline. All the patients will be treated by means of non surgical periodontal therapy on a quadrant protocol including oral hygiene instructions and motivations and subgingival instrumentation in four successive visits. 6 weeks after the last visit, the clinical parameters will be registered again.

Clinical Parameters:

Periodontal condition of each patient will be evaluated through the collection of the following parameters:

* Full-Mouth Bleeding score (FMBS): presence/absence of bleeding on probing using a periodontal probe on each surface of the tooth (six sites per tooth), calculated in percentage for all the examined teeth.
* Full-Mouth Plaque Score (FMPS): presence/absence of plaque using a periodontal probe on each surface of the tooth (six sites per tooth), calculated in percentage for all the examined teeth.
* Probing Depth (PD): measured for each surface of the tooth (six sites per tooth) using a periodontal probe, measured as the distance between the cementoenamel junction (CEJ) and the depth of the pocket.
* Gingival recession (Rec): measured for each surface of the tooth (six sites per tooth) using a periodontal probe, measured as the distance between the cementoenamel junction (CEJ) and the free gingival margin.
* Clinical attachment level (CAL): The sum of PD and Rec.

Psychologic Test:

The Stress condition of each patient will be assessed by a Psychologist using:

PSS is a 10-items self-report questionnaire that measure the degree to which situations in one's life are appraised as stressful. The PSS is scored on a 5-point scale (never, almost never, sometimes, fairly often and very often). PSS norms are available from a sample of the USA collected by Cohen & Williamson (1988). The mean level for men was 12.1 (S.D. 5.9) and for women 13.7 (S.D. 6.6).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Periodontitis stage III/IV according to the new classification (2018);
* Presence of at least 14 teeth, with a minimum of 10 sites with PD at least > 5 mm and radiographic evidence of alveolar bone loss.
* Written informed consent

Exclusion Criteria:

* Smokers > 10 cig/die
* Patients with orthodontic appliances;
* Pregnant or lactating women;
* Individuals who have received periodontal treatment in the 6 months prior to recruitment;
* Patients with systemic diseases that could interfere the clinical response to periodontal treatment (i.e. diabetes);
* Subjects under treatment with antibiotics, steroidal and/or non-steroidal anti-inflammatory medication 3 weeks prior to the visit and patients treated with antiepileptic drugs.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Full Mouth Bleeding Score FMBS% (0 - 100 % with higher percentage indicating worse status) | Baseline and 6 weeks after the completion of the therapy.
  Percentage of full mouth bleeding sites after probing considering 6 sites for each tooth.

SECONDARY OUTCOMES:
Change in Full Mouth Plaque Score FMPS% (0 - 100 % with higher percentage indicating worse status) | Baseline and 6 weeks after the completion of the therapy.
  Percentage of full mouth plaque score considering 6 sited for each tooth.
Change in Probing Pocket Depth PD (0 - 15mm with higher values indicating worse outcomes. | Baseline and 6 weeks after the completion of the therapy.
  The distance between the cementoenamel junction (CEJ) and the base of the pocket.
Change in Gingival Recession Rec (0 - 15mm with higher values indicating worse outcomes. | Baseline and 6 weeks after the completion of the therapy.
  The distance between the cementoenamel junction (CEJ) and the free gingival margin
Change in Clinical Attachment Level CAL (0 - 15mm with higher values indicating worse outcomes. | Baseline and 6 weeks after the completion of the therapy.
  The sum of Probing pocket depth (PD) and Recession (Rec)

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romano F, Bebars A, Ortu V, Bottone M, Giraudi M, Mariani GM, Baima G, Aimetti M. Effect of psychosocial stress and coping strategies on non-surgical periodontal therapy in patients with generalized stage III/IV periodontitis: a longitudinal intervention study. Clin Oral Investig. 2023 Jul;27(7):3479-3487. doi: 10.1007/s00784-023-04956-w. Epub 2023 Mar 24. PMID 36961591